CLINICAL TRIAL: NCT03091166
Title: The Effect of Prophylactic Dexmedetomidine Administration on the Outcome in Patients Undergoing Surgery With Cardiopulmonary Bypass
Brief Title: Effect of Perioperative Dexmedetomidine Administration on Outcome in Cardiac Surgery Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Moscow Regional Research and Clinical Institute (MONIKI) (Other Government)
Responsible Party: Principal Investigator, Oleg A. Grebenchikov, senior researcher, Moscow Regional Research and Clinical Institute (MONIKI)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PD-CS-2016
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Patient Outcome Assessment
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine (Active Comparator)
  Interventions: Drug: Dexmedetomidine
- No Dexmedetomidine (No Intervention)

INTERVENTIONS:
Drug: Dexmedetomidine
  Other Names: Dexdor
  Arms: Dexmedetomidine

SUMMARY:
Investigation of effect of perioperative Dexmedetomedine administration on mortality, length of ICU and hospital stay, delirium onset, major adverse cardiac and cerebrovascular events, acute kidney injury in cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed agreement
* Elective surgery
* Use of CPB

Exclusion Criteria:

* Previous prolonged immobilization
* Reoperation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2016-12; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
30DM | 30 days after surgery
  30-day mortality
Delirium | 30 days after surgery
  Postoperative delirium

SECONDARY OUTCOMES:
VIS | 5 days after surgery
  Vasoactive- Inotropic Score
MACCE | 30 days after surgery
  Major adverse cardiac and cerebrovascular events
Subsyndromal delirium | 30 days after surgery
  Subsyndromal postoperative delirium
AKI | 7 days after surgery
  Acute kidney injury
ICU-LOS | 7 days after surgery
  Length of ICU stay
H-LOS | 30 days after surgery
  Hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Valery Likhvantsev, Professor, Principal Investigator — Moscow Regional Clinical and Research Institute, Moscow, Russia
Locations (1):
- Moscow Regional Research and Clinical Institute Moniki n.a. M.F. Vladimirskiy, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No